CLINICAL TRIAL: NCT00292500
Title: Efficacy of Automated Distal Vascular Anastomosis in Coronary Surgery: Phase II
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Cardica has terminated the development of the product for Business Reason.
Sponsor: Cardica, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP2004-06
Record Dates: First submitted 2006-02-14; First posted 2006-02-16 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Coronary Artery Disease
Keywords: CABG, anastomotic device; myocardial revascularization
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- C-Port (No Intervention): Automated distal anastomotic device
  Interventions: Device: Automated distal anastomotic device

INTERVENTIONS:
Device: Automated distal anastomotic device — CABG
  Other Names: C-Port xA Distal Anastomosis System

SUMMARY:
This evaluation is designed to evaluate the feasibility of using an automated distal coronary anastomotic to facilitate grafting of the left internal mammary artery to the left anterio descending coronary artery during myocardial revascularization in patients with coronary artery disease requiring surgical intervention. The study is designed to assess the ability to compare the patency of grafts created using an automated device versus hand-sewn grafts of the same vessels in the same patient population.

DETAILED DESCRIPTION:
Evaluation of automated distal anastomotic device as a surrogate for hand-sewn grafts for completion of arterial conduit anastomosis between the Left Internal Mammary Artery and Left Anterior Descending Artery among patients with coronary artery disease requiring surgical revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 85 years (inclusive)
* Diagnostically confirmed coronary disease
* Ejection fraction > 30%
* Tolerate contrast media
* Acceptable LIMA (conduit) and LAD (target)for grafting
* Life expectancy > 1 year

Exclusion Criteria:

* Refusal to give informed consent
* Unable to meet study travel and general health requirements
* Pregnancy
* Previous cardiac surgery
* NYHA Class IV
* Preoperative need for IABP
* Acute or chronic dialysis (creatinine > 200mmolor 2.3 mg/dL) within 30 days of surgery
* Acute or suspected systemic infection
* Need for ongoing immunosuppressive therapy
* Recent history (<2 weeks) of CVA
* Aspirin allergy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2006-01; Primary Completion 2008-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Coronary patency of index graft at the sixth post-operative month | 6 months post-op

SECONDARY OUTCOMES:
Establish preliminary safety profile | 6 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Jan Gummert, MD, Principal Investigator — Herzzentrum Leipzig Gmbh
Locations (1):
- Klinik für Herzchirurgie, Leipzig, Germany